CLINICAL TRIAL: NCT01950897
Title: Establishment of Phenotypic Profiles of Muscular Dystrophies for Understanding Disease Progression, Diagnosis and Development of New Therapies
Brief Title: Muscle Tissue Bank for Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: CHS-Neurology-MD Muscle Tissue
Record Dates: First submitted 2013-03-30; First posted 2013-09-26 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2019-12

CONDITIONS: Muscular Dystrophies; Muscular Dystrophy
Keywords: muscular dystrophies; muscular dystrophy
MeSH Terms: conditions — Muscular Dystrophies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — skeletal muscle tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- subjects dx'd clinically w/ muscular dystrophy: subjects with muscular dystrophy from whom muscle samples are obtained for clinical diagnosis or for any other medical purpose
- normal controls: subjects who do not have muscular dystrophy and from whom muscle samples are obtained for any medical purpose

SUMMARY:
This protocol proposes to establish gene expression profiles of muscular dystrophies for correct diagnosis and for development of experimental therapies for these diseases.

DETAILED DESCRIPTION:
Muscular dystrophies are caused by mutations in more than 30 genes, some of them remaining to be identified. Phenotypically, it is known that one specific mutation can affect the expression of several other proteins causing difficulty in diagnosis. Correct genotyping is essential for diagnosis, prognosis and treatment, and relies on a complexed analysis of muscle tissues for phenotype profiles. Our research aims to understand how different gene mutations affect expression of other genes via muscle biopsy samples and establishment of phenotypic profiles for correct diagnosis of individual patients. Establishment of such information will be critical for understanding the progression of different muscular dystrophies and to devise new experimental therapies. This research will also provide vital clues for finding new genes involved in the disease process. Muscle samples may also be used to establish cell cultures for testing drugs and new therapies relevant to the treatment of the muscular dystrophies.

ELIGIBILITY:
Inclusion Criteria:

* subjects with or without muscular dystrophy who will be undergoing a diagnostic or therapeutic procedure that involves the removal of a sample of skeletal muscle tissue.
* subjects with or without muscular dystrophy who have had a previous skeletal muscle biopsy performed and where a portion of the muscle sample remains in medical storage are also eligible for this study.

Exclusion Criteria:

* Under age 6

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to the Carolinas Medical Center (CMC) Department of Neurology who meet study criteria.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2005-08-24 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2015-06-09 (Actual)

PRIMARY OUTCOMES:
Immunohistochemistry for protein expression profiling of skeletal muscle tissue; initial analysis will be qualitative (positive or negative) or semi-quantitative (strong, moderate, weak or negative) | Data will be analyzed at one year.
  Samples of MD subjects will be compared to samples of non-muscular dystrophy subjects (i.e. control samples).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin R Brooks, MD, Principal Investigator — Medical Director, Carolinas Neuromuscular/ALS-MDA Center, CMC
Locations (1):
- Carolinas Medical Center - Dept of Neurology, Charlotte, North Carolina, United States